CLINICAL TRIAL: NCT06173544
Title: HIV Engagement and Adolescent Depression Support (HEADS-UP)
Acronym: HEADS-UP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: RTI International (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23-2439; R34MH130232 (NIH)
Record Dates: First submitted 2023-12-07; First posted 2023-12-15 (Actual); Last update posted 2025-05-26 (Actual); Status verified 2025-05

CONDITIONS: Depression; Anxiety; Adolescent Behavior; HIV Infections; Immune System Diseases
MeSH Terms: conditions — Depression; Anxiety Disorders; Adolescent Behavior; HIV Infections; Immune System Diseases | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Three-Arm Individually Randomized Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Standard of Care (SOC) (Active Comparator): 35 adolescents living with HIV seeking HIV care at participating clinics in Lilongwe, Malawi will be enrolled in this study arm during study recruitment. Enhanced usual care will include general training of the HIV providers and clinics about common mental disorder (CMD) identification and management, and feedback to the HIV provider of the status of their enrolled patient to allow follow-up per the clinic's standard care. Enhanced usual care will included a mental health evaluation provided by a rained study nurse; brief supportive counseling; information, education, and support on depression; and (if indicated) facilitation of referral to the clinic's psychiatric nurse or mental health clinic or to the tertiary care hospital.
  Interventions: Behavioral: Standard of Care (SOC)
- Adapted Friendship Bench (AFB) (Experimental): 35 adolescents living with HIV seeking HIV care at participating clinics in Lilongwe, Malawi will be enrolled in this study arm during study recruitment. Individuals enrolled in this arm will receive 6 weekly counseling sessions per the AFB protocol.
  Interventions: Behavioral: Adapted Friendship Bench (AFB)
- Enhanced Friendship Bench (EFB) (Experimental): 35 adolescents living with HIV seeking HIV care at participating clinics in Lilongwe, Malawi will be enrolled in this study arm during study recruitment. Individuals enrolled in this arm will receive 6 weekly counseling sessions and peer support per the EFB protocol.
  Interventions: Behavioral: Enhanced Friendship Bench (EFB)

INTERVENTIONS:
Behavioral: Standard of Care (SOC) — Participants randomized to this arm will received enhanced standard of care.
  Arms: Standard of Care (SOC)
Behavioral: Adapted Friendship Bench (AFB) — Participants randomized to this arm will receive the Adapted Friendship Bench protocol delivered by a trained counselor.
  Arms: Adapted Friendship Bench (AFB)
Behavioral: Enhanced Friendship Bench (EFB) — Participants randomized to this arm will receive the Enhanced Friendship Bench protocol delivered by a trained counselor and a peer supporter.
  Arms: Enhanced Friendship Bench (EFB)

SUMMARY:
This pilot study will individually randomize 105 adolescents living with HIV 1:1:1 to standard of care, adapted intervention, or enhanced intervention. The intervention is called the Friendship Bench Intervention is a counseling intervention for depression and engagement in HIV care.

DETAILED DESCRIPTION:
Sub-Saharan Africa is home to the largest population of adolescents living with HIV (ALWH). Engaging ALWH in HIV care is challenging and reflected in lower rates of viral suppression and higher rates of loss to follow-up as compared to adults in the region. Depression has been identified as a significant barrier to initiating and remaining in HIV care. Indeed, this is the case for ALWH in Malawi where estimates of viral suppression range from 40%-78% and estimates of depression range from 18-26%. Resource-appropriate interventions that improve depression and address engagement in HIV care for ALWH are urgently needed.

The Friendship Bench (FB) is an evidence-based depression counseling intervention delivered by trained, supervised lay health workers. It is proven to reduce depression in the general population in low-resource settings but has not been adapted to be youth-friendly or enhanced with peer support to facilitate engagement in HIV care among ALWH. FB is based on problem-solving therapy, which offers an ideal framework for youth-friendly adaption and integration of retention peer support into a proven depression treatment model.

The long-term goal of the study team is to adapt, test, and scale up resource-appropriate interventions to reduce depression and improve engagement in HIV care amongst ALWH. The specific aims are: 1) to conduct formative research for youth-friendly adaptation and peer support enhancement of FB; 2) to adapt the evidence-based FB protocol to meet the developmental and contextual needs of ALWH and enhance this adapted FB protocol with peer support to facilitate HIV care engagement among ALWH; and 3) to determine the feasibility, fidelity, and acceptability of the Adapted and Enhanced FB protocols to improve depression and engagement in HIV care among ALWH. For the latter, a 3-arm individually randomized pilot study will be conducted to compare the adapted FB and the enhanced FB to standard care. The proposed aims pave the way for a R01 application to test the adapted and enhanced Friendship Bench interventions in a cluster randomized controlled trial and represent an important step forward towards improving depression among ALWH.

ELIGIBILITY:
Inclusion Criteria:

* age 13-18
* diagnosed with HIV (vertically or horizontally)
* scored ≥ 13 on the self-reported and previously used BDI-II
* living in the clinic's catchment area with intention to remain for > 1 year
* willing to provide consent (age 18 or 16-17 years old and married (emancipated minors per Malawi law) or assent with parental consent (age 13-17)

Exclusion Criteria:

* Less than 13 or greater than 18 years of age

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 105 (Estimated)
Dates: Start 2024-07-06 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Recruitment Rate (Intervention Feasibility) | Baseline
  This measure is the ability to successfully enroll adolescents living with HIV (ALWH) in the pilot trial. Feasibility will be evaluated by measuring the recruitment rate (number of patients approached in order to accrue the final sample).
Number of participants retained in the study (Intervention Feasibility) | 12 months
  This measure of feasibility will be measured as the ability to retain adolescents living with HIV (ALWH) in the pilot trial. Feasibility will be evaluated by measuring the number of participants retained in the study (number of patients enrolled at baseline who are still enrolled in the trial), through study completion.
Proportion of sessions attended (Intervention Feasibility) | 12 Months
  The number of sessions attended by participants out of total number of sessions offered.
Number of sessions meeting Fidelity Threshold (Intervention Fidelity) | 12 Months
  Fidelity to content for sessions will be assessed by a member of the research team using a checklist of intervention characteristics. Intervention fidelity will be measured as the total number of sessions meeting or exceeding expectations for at least 80% of the total number of fidelity checklist items assessed per session.
Overall Satisfaction among Participants (Intervention Acceptability) | 12 Months
  Acceptability will be assessed through brief exit interviews with a sample of adolescents living with HIV (ALWH), all study staff, and supervisors. Exit interviews will assess how easy the intervention was to participate in or deliver, the perceived usefulness of the intervention, suggestions for improvement, and will explore contextual factors that impeded or facilitated implementation.
  Intervention acceptability will be measured as the number of participants who were either very satisfied or somewhat satisfied with the intervention. Satisfaction will be measured on a 4-point Likert scale-- 1 indicates high satisfaction and 4 indicates high dissatisfaction.

SECONDARY OUTCOMES:
Change in depression symptoms from baseline | Baseline,12 months
  Change in depression symptoms from baseline will be evaluated using Beck's Depression Inventory (BDI-II). The Beck Depression Inventory (BDI-II) is a 21-item patient self-report measure of the severity of depression. Each item is rated on a 4-point scale ranging from 0 to 3. The minimum total score is zero and the maximum total score is 63. A total score of 0-13 is considered nondepressed, 14-19 represents mild depression, 20-28 represents moderate depression, and 29-63 represents severe depression. Lower scores represent better outcomes. Scores reported are change in symptoms relative to baseline.
Number of adolescents living with HIV who attended at least one appointment per quarter | 12 months
  Number of adolescents living with HIV who attended at least one appointment per quarter.
Number of Participants Achieving HIV Viral Suppression | 12 months
  Number of participants achieving HIV viral suppression at 12 months (HIV RNA < 1000 copies/mL).

CONTACTS AND LOCATIONS:
Overall Officials: Bradley N Gaynes, MD, Principal Investigator — University of North Carolina, Chapel Hill; Nivedita L Bhushan, PhD, Principal Investigator — RTI International
Locations (5):
- Malawi (5):
  - Area 18 Health Centre, Lilongwe
  - Area 25 Health Centre, Lilongwe
  - Kawale Health Centre, Lilongwe
  - Lighthouse Health Centre, Lilongwe
  - UNC Project Malawi, Lilongwe

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with the University of North Carolina at Chapel Hill (UNC).
Time Frame: beginning 9 and continuing for 36 months after publication
Access Criteria: Investigator has approved IRB, IEC, or REB and an executed data use/sharing agreement with UNC.

REFERENCES:
- [Derived] Dao TTD, Gaynes BN, Pence BW, Mphonda SM, Kulisewa K, Udedi M, Stockton MA, Kramer J, Waddell KG, Faidas M, Mortensen H, Bhushan NL. Friendship Bench intervention to address depression and improve HIV care engagement among adolescents living with HIV in Malawi: Study protocol for a pilot randomized controlled trial. PLoS One. 2025 Mar 19;20(3):e0302666. doi: 10.1371/journal.pone.0302666. eCollection 2025. PMID 40106412